CLINICAL TRIAL: NCT01058174
Title: Randomized, Open Label, Non-inferiority Study of Micafungin Versus Standard Care for the Prevention of Invasive Fungal Disease in High Risk Liver Transplant Recipients
Brief Title: Liver Transplant European Study Into the Prevention of Fungal Infection
Acronym: TENPIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9463-EC-0001; 2008-005214-49 (EudraCT Number)
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Liver Transplantation; Mycoses
Keywords: Prophylaxis; Liver transplantation; Invasive Fungal Infection; Micafungin; Prevention; Mycoses
MeSH Terms: conditions — Mycoses; Invasive Fungal Infections | interventions — Micafungin; Fluconazole; liposomal amphotericin B; Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- micafungin (Experimental): intravenous infusion
  Interventions: Drug: micafungin
- standard care (Active Comparator): intravenous infusion
  Interventions: Drug: fluconazole; Drug: liposomal amphotericin B; Drug: caspofungin

INTERVENTIONS:
Drug: micafungin — intravenous infusion
  Other Names: Mycamine
  Arms: micafungin
Drug: fluconazole — intravenous infusion
  Other Names: Diflucan
  Arms: standard care
Drug: liposomal amphotericin B — intravenous infusion
  Other Names: AmBisome
  Arms: standard care
Drug: caspofungin — intravenous infusion
  Other Names: Cancidas
  Arms: standard care

SUMMARY:
Prevention of invasive fungal infection in high risk patients following liver transplant.

DETAILED DESCRIPTION:
After receiving liver transplant, subjects will be randomized to one of the two treatment arms.

Study drugs will be administered for a period of 21 days, or until hospital discharge, whichever occurs first.

Additionally, mortality data will be collected at the Long-term Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing orthotopic whole or split liver allograft transplantation
* Patients at 'high risk' of invasive fungal infection due to the presence of at least one of the following risk factors:

  * Re-transplantation
  * Acute liver failure
  * Pre- or post-operative renal impairment (defined as creatinine clearance ≤40 ml/min) or need for renal replacement therapy
  * Admission to Intensive Care Unit (ICU) for greater than 48 hours prior to liver transplant
  * Re-operation (abdominal surgery) within 5 days of liver transplant
  * Presence of choledocojejunostomy
  * Perioperative colonization with fungi, defined as two or more positive clinical site surveillance cultures for Candida spp., obtained within 96 hours before or after liver transplant
  * Need for prolonged mechanical ventilation for greater than 48 hours following liver transplant
  * Transfusion intraoperatively of 20 or more units of cellular blood products
* Female subject of childbearing potential must have a negative urine or serum pregnancy test prior to randomization and must agree to maintain effective birth control during the study

Exclusion Criteria:

* Any systemic antifungal therapy (excluding fluconazole or oral nystatin for a maximum of 7 days) within 14 days prior to randomization
* Evidence of documented ('proven' or 'probable') or suspected ('possible') IFD (according to the EORTC/MSG criteria)
* Allergy, hypersensitivity, or any serious reaction to an echinocandin antifungal, or any of the study drugs or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2009-12-15 (Actual); Primary Completion 2012-05-03 (Actual); Study Completion 2012-05-03 (Actual)

PRIMARY OUTCOMES:
'Clinical success' at the End of Prophylaxis as assessed by the Independent Data Review Board (IDRB). | up to 21 days

SECONDARY OUTCOMES:
Absence of a 'proven' or 'probable' Invasive Fungal Disease (IFD) at the End of Study as assessed by the IDRB | 3 months
Absence of 'proven' or 'probable' IFD at the End of Prophylaxis and at the End of Study as assessed by the Investigator | up to 21 days & 3 months
Time to 'proven' or 'probable' IFD | up to 3 months
Fungal free survival at the End of Study and at the end of Long-term Follow-up | 3 months & 6 months
Incidence of superficial fungal infection and colonization at the End of Prophylaxis as compared to Baseline | up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe Ltd.
Locations (33):
- Innsbruck, Austria
- Belgium (3):
  - Antwerp
  - Brussels
  - Ghent
- France (4):
  - Paris, Villejuif Cedex
  - Clichy
  - Paris
  - Toulouse
- Germany (4):
  - Berlin
  - Hamburg
  - Hanover
  - Heidelberg
- Budapest, Hungary
- Dublin, Ireland
- Italy (4):
  - Milan
  - Padua
  - Torino
  - Udine
- Portugal (2):
  - Coimbra
  - Porto
- Bucharest, Romania
- Russia (2):
  - Moscow
  - Saint Petersburg
- Riyadh, Saudi Arabia
- Spain (6):
  - Santiago de Compostela, A Coruna
  - Barakald, Vicaya
  - Barcelona
  - Córdoba
  - Madrid
  - Valencia
- Stockholm, Sweden
- United Kingdom (2):
  - Birmingham
  - London

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Saliba F, Pascher A, Cointault O, Laterre PF, Cervera C, De Waele JJ, Cillo U, Langer RM, Lugano M, Goran-Ericzon B, Phillips S, Tweddle L, Karas A, Brown M, Fischer L; TENPIN (Liver Transplant European Study Into the Prevention of Fungal Infection) Investigators; TENPIN Liver Transplant European Study Into the Prevention of Fungal Infection Investigators. Randomized trial of micafungin for the prevention of invasive fungal infection in high-risk liver transplant recipients. Clin Infect Dis. 2015 Apr 1;60(7):997-1006. doi: 10.1093/cid/ciu1128. Epub 2014 Dec 17. PMID 25520332
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=50